CLINICAL TRIAL: NCT02192008
Title: Investigating the Mechanisms and Determinants of Systemic and Mucosal Immunity to Salmonella Typhi and Salmonella Paratyphi A in naïve and Previously Exposed Individuals - A Challenge and Rechallenge Study
Brief Title: Investigating Enteric Fever - Salmonella Typhi and Paratyphi Challenge Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: University of Liverpool (Other); Brigham and Women's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: OVG 2014/01
Record Dates: First submitted 2014-07-01; First posted 2014-07-16 (Estimated); Last update posted 2022-06-02 (Actual); Status verified 2021-01

CONDITIONS: Typhoid Fever; Paratyphoid Fever
Keywords: Challenge; Re-challenge; Controlled Infection; Enteric fever
MeSH Terms: conditions — Typhoid Fever; Paratyphoid Fever

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Part A (Active Comparator): Cohort naive to typhoidal Salmonella challenged with either S. Typhi or S. Paratyphi
  Interventions: Biological: Salmonella Typhi; Biological: Salmonella Paratyphi
- Part B (Active Comparator): Cohort previously challenged with S. Typhi or Paratyphi re-challenged with either S. Typhi or S. Paratyphi.
  Interventions: Biological: Salmonella Typhi; Biological: Salmonella Paratyphi

INTERVENTIONS:
Biological: Salmonella Typhi
Biological: Salmonella Paratyphi

SUMMARY:
Enteric fever, an infection characterised by diarrhoea and rash, is most often caused by a bacteria called Salmonella enterica. After ingesting contaminated food or drink, the Salmonellae travel first to the gut, then the bloodstream, from where they can infect other parts of the body. Antibiotics are used to kill the bacteria, but with increasing rates of antibiotic resistance, this treatment is becoming less effective.

Two Salmonella variants, Typhi and Paratyphi, cause over 30 million cases of enteric fever and more than 200,000 deaths per year, mostly in developing countries. While improved hygiene and sanitation should eventually eliminate enteric fever, reduction of the disease burden in the medium term is achievable through effective vaccination.

Vaccines likely to be available for mass vaccination are effective only against those Salmonella strains that bear the Vi polysaccharide capsule protein. Strains that do not have these capsule proteins, or have no capsule, will not be affected by vaccination and could 'fill' the space vacated by the capsulated strains. Indeed, enteric fever caused by S. Paratyphi A which does not carry the Vi protein, has risen during the past decade and accounts for more than half of all cases in some areas. Thus it is important that effective vaccines are available to protect against infection by both capsulated and noncapsulated Salmonella enterica. To develop such vaccines, we need a complete understanding of the human immune response to both types, including the contribution of immunity in the gut and the bloodstream, immune response to bacterial surface proteins, and the role of antibodies. How much cross-protection there is between the types of typhoidal Salmonellae after natural infection or vaccination is not known, but this is critical to vaccine development.

This project aims to fill in the knowledge gaps highlighted, by fully characterising the infection process and immune response in enteric fever.

DETAILED DESCRIPTION:
There are two main groups in this study. Firstly a group of 40 to 60 volunteers recruited from the community and not previously exposed to typhoidal Salmonella (part A); secondly a group of 20 to 60 volunteers from participants of previous challenge studies conducted by the Oxford Vaccine Group (part B).

Participants in part A and B will be randomly allocated one-to-one to have either S. Typhi or S. Paratyphi. The dose of bacteria has been determined by previous challenge studies to give an attack rate of 60 to 75% in individuals naive to typhoidal Salmonella. The bacteria is then ingested as a drink with a bicarbonate buffer ('the challenge').

In addition to these two groups, a preliminary study involving 3 to 10 participants to act as 'negative controls' will be performed. They will ingest the bicarbonate drink but not be given S. Typhi or S. Paratyphi. This group is not randomised with part A or B, and is unblinded i.e. the participant will be aware that they are not drinking typhoidal Salmonella. The participants will have all the same procedures and investigations as those in part A and B, including endoscopy with biopsies, daily visits during the two week intensive phase, and a course of antibiotics.

Prior to challenge, participants (from parts A, B and negative control group) will undergo endoscopy and tissue biopsies of the gut lining. This procedure will be repeated after the intensive phase and completion of a two week course of antibiotics.

After challenge, participants will be reviewed daily for at least 14 days by study investigators. Samples of blood, stool, saliva and urine will be collected. Participants diagnosed with enteric fever will be treated immediately with antibiotics and samples will be taken as per the protocol. The participants who do not meet criteria for enteric fever will be treated with antibiotics on Day 14.

Enteric fever is diagnosed if any of the following apply:

1. A positive blood culture for S. Typhi or Paratyphi from 72 hours post-challenge,
2. a positive blood culture for S. Typhi or Paratyphi within 72 hours post-challenge, with one or more signs/symptoms of enteric fever,
3. persistent positive blood cultures (two or more blood cultures taken at least 4 hours apart) for S. Typhi or Paratyphi within 72 hours postchallenge, or
4. oral temperature ≥ to 38°C persisting for 12 hours.

A proportion of participants from Part A and B will be offered the optional procedures of enteric string tests (also called Enterotest) and/or Wireless Video Capsule Endoscopies (WCE). Participants consenting to these procedures will be selected sequentially until the quota has been filled for each group.

ELIGIBILITY:
Inclusion Criteria:

* In good health as determined by medical history, physical examination and clinical judgment of the investigators.
* Agree (in the Investigator's opinion) to comply with all study requirements, including capacity to adhere to good personal hygiene and infection control precautions.
* Agree to allow his or her General Practitioner (and/or Consultant if appropriate), to be notified of participation in the study.
* Agree to allow Public Health England to be informed of their participation in the study .
* Agree to give his or her close household contacts written information informing them of the participants' involvement in the study and offering them voluntary screening for S. Typhi or S. Paratyphi carriage.
* Agree to have 24-hour contact with study staff during the four weeks post challenge and are able to ensure that they are contactable by mobile phone for the duration of the challenge period until antibiotic completion.
* Have internet access to allow completion of the e-diary and real-time safety monitoring.
* Agree to avoid antipyretic/anti-inflammatory treatment until advised by a study doctor or until at least 14 days after challenge.
* Willing to undergo endoscopy and biopsy.

Exclusion Criteria:

* History of significant organ/system disease that could interfere with study conduct or completion.
* Have any known or suspected impairment of immune function, alteration of immune function, or prior immune exposure that may alter immune function.
* Moderate or severe depression or anxiety as classified by the Hospital Anxiety and Depression Score at screening or challenge that is deemed clinically significant by the study investigators.
* Weight 50kg or less.
* Presence of implants or prosthesis.
* Have previously received any typhoid vaccine
* Any contraindication to elective upper GI endoscopy.
* More than one non-study related upper GI endoscopy within the last year.
* Anyone taking long-term medication that may affect symptom reporting or interpretation of the study results.
* Contra-indication to taking ciprofloxacin, azithromycin, trimethoprim/ sulfamethoxazole and/or beta lactam antibiotics.
* Female participants who are pregnant or lactating.
* Female participants who are unwilling to ensure that they or their partner use effective contraception one month prior to challenge and continue to do so until two negative stool samples, a minimum of three weeks after completion of antibiotic treatment, have been obtained.
* Full-time, part-time or voluntary occupations involving clinical or social work with direct contact with young children (defined as those attending pre-school groups or nursery or aged under 2 years); clinical or social work with direct contact with highly susceptible patients or persons in whom typhoid or paratyphoid infection would have particularly serious consequences e.g. the elderly or infirm.
* Full time, part time or voluntary occupations involving commercial food handling.
* Close household contact with young children (defined as those attending pre-school groups, nursery or those aged less than 2 years), individual(s) who is (are) immunocompromised, scheduled elective surgery or other procedures requiring general anaesthesia during the study period.
* Participants who have participated in another research study involving an investigational product that might affect risk of typhoid or paratyphoid infection or compromise the integrity of the study within the 30 days prior to enrolment .
* Detection of any significantly abnormal results from screening investigations.
* Inability to comply with any of the study requirements.
* Any other social, psychological or health issues which, in the opinion of the study investigator, may put the participants or their contacts at risk because of participation in the study, adversely affect the interpretation of the primary endpoint data, or impair the participant's ability to participate in the study.
* Having been resident in an enteric fever endemic country for six months or more.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 125 (Actual)
Dates: Start 2014-12; Primary Completion 2018-09-22 (Actual); Study Completion 2022-05-26 (Actual)

PRIMARY OUTCOMES:
Measure the attack rate after challenge with S. Typhi or S. Paratyphi A in naïve and previously challenged individuals. | 12 months
  Based on clinical and/or microbiological proven enteric fever infection.

SECONDARY OUTCOMES:
To describe the human clinical response to S. Typhi or S. Paratyphi A in antigen-naïve and previously challenged individuals. | 12 months
  The clinical response after challenge or re-challenge using participant symptom profiles, laboratory parameters (including inflammatory markers, blood count, liver function tests and microbiological culture results) will be used.
To describe the characteristics of bacterial dynamics after challenge in naïve and previously exposed individuals, including onset and duration of bacteraemia, bacterial burden at diagnosis, bacterial burden in enteric fluid, and stool shedding. | 12 months
  Microbiological culture (qualitative and quantitative) and polymerase chain reaction to detect and characterise S. Typhi or S. Paratyphi A in blood, stool and enteric fluid.
To determine the gut luminal mucosal response to challenge with S. Typhi and S. Paratyphi. | 12 months
  Mucosal inflammation as determined by (1) macroscopic appearance of mucosal inflammation as seen on endoscopy and wireless video capsule endoscopy (judged by experienced endoscopists), (2) inflammatory markers such as calprotectin and lactoferrin performed on stool and duodenal secretions.
To describe the human immune response to challenge or re-challenge, including the innate, humoral, cell-mediated and mucosal responses. | 12 months
  Assessed by immunological laboratory assays including quantitative and functional assays of the humoral (e.g. ELISA, enzyme-linked immunospot, serum bactericidal assay and opsonophagocytosis assay), mucosal (secretory immunoglobulin A measurement), and cell-mediated (multi-chromatic flow cytometry, mass cytometry, cytokine measurement) immune response.
Determine host genetic features influencing: • clinical manifestations of challenge with typhi/paratyphi • alteration of those responses through epigenetic changes • and control of gene and protein expression. | 12 months
  Assessed by laboratory and high-throughput assays including:
  * measurement of baseline genetic susceptibility factors by whole genome sequencing
  * the transcriptional response to challenge and infection
  * detection of translated proteins by mass spectrometry (CyTOF).

OTHER OUTCOMES:
Exploratory immunology to investigate the innate, humoral, cell-mediated and mucosal responses to challenge with S. Typhi or S. Paratyphi A in naïve and previously challenged individuals. | 5 years
  Novel assays performed on peripheral blood, faeces, urine, saliva and mucosal biopsies, including assays for CD1 and MR1 restricted T cell responses and whole blood and peripheral blood mononuclear cell (PBMC) killing assays.
To investigate how the human microbiome influences and interacts with a challenge of S. Typhi or S. Paratyphi A | 5 years
  Samples of stool and enteric fluid to measure the constituent microbiological flora by assays such as pyrosequencing and related metagenomic studies.
Investigate new molecular techniques for detection of S. Typhi and/or S. Paratyphi in clinical samples. | 5 years
  Use of novel methodologies to prepare bacterial DNA/RNA and development of sensitive quantitative and qualitative PCR assays for blood, stool and duodenal secretions.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Pollard, FRCPCH, PhD, Principal Investigator — University of Oxford
Locations (1):
- Oxford Vaccine Group, Oxford, Oxfordshire, United Kingdom

REFERENCES:
- [Background] Gibani MM, Jin C, Shrestha S, Moore M, Norman L, Voysey M, Jones E, Blackwell L, Thomaides-Brears H, Hill J, Blohmke CJ, Dobinson HC, Baker P, Jones C, Campbell D, Mujadidi YF, Plested E, Preciado-Llanes L, Napolitani G, Simmons A, Gordon MA, Angus B, Darton TC, Cerundulo V, Pollard AJ. Homologous and heterologous re-challenge with Salmonella Typhi and Salmonella Paratyphi A in a randomised controlled human infection model. PLoS Negl Trop Dis. 2020 Oct 20;14(10):e0008783. doi: 10.1371/journal.pntd.0008783. eCollection 2020 Oct. PMID 33079959
- [Derived] Jin C, Gibani MM, Pennington SH, Liu X, Ardrey A, Aljayyoussi G, Moore M, Angus B, Parry CM, Biagini GA, Feasey NA, Pollard AJ. Treatment responses to Azithromycin and Ciprofloxacin in uncomplicated Salmonella Typhi infection: A comparison of Clinical and Microbiological Data from a Controlled Human Infection Model. PLoS Negl Trop Dis. 2019 Dec 26;13(12):e0007955. doi: 10.1371/journal.pntd.0007955. eCollection 2019 Dec. PMID 31877141
- See also: Homologous and heterologous re-challenge with Salmonella Typhi and Salmonella Paratyphi A in a randomised controlled human infection model — https://journals.plos.org/plosntds/article?id=10.1371/journal.pntd.0008783
- See also: Related Info — http://www.nature.com/articles/s41590-018-0133-z
- See also: Related Info — http://www.nature.com/articles/s41467-017-02540-x